CLINICAL TRIAL: NCT07209917
Title: Secondary Cervical Cancer Prevention of Vulnerable Women With Human Papillomavirus (HPV) and Human Immunodeficiency Virus (HIV) Co-infection in India
Brief Title: Secondary Cervical Cancer Prevention of Vulnerable Women With HPV and HIV Co-infection in India
Acronym: ASHA-Health II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, San Francisco (Other); National Institute of Mental Health and Neuro Sciences (NIMHANS) (Unknown)
Responsible Party: Principal Investigator, Adeline Nyamathi, Distinguished Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2988-2962; 1R01CA285063-01 (NIH)
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Human Papillomavirus (HPV) Infection; Human Immunodeficiency Virus (HIV) Infection
Keywords: Cervical Cancer Prevention; HPV-HIV Co-Infection; ASHA-Nutrition
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections; Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: In Phase 2 (mos 12 - 41) + follow-ups, the investigators will conduct a two-arm parallel-group RCT among 420 W-Co-V who are cared for at ART centers in Bangalore and northern Karnataka. Participants will be allocated to the ASHA-Health and SOC+ study arms through individual randomization in a 1:1 ratio prior to study enrollment. A cohort of 84 women (42 per group) will be enrolled every six months.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASHA-Health (Experimental): The ASHA-Health program will include: 1) 8 group sessions, led by the nurse, and inclusive of other experts (such as HPV/HIV physician, nutritionist, psychologist) to provide the group classes for each cohort of 42 W-Co-V in the program, covering content about staying healthy, taking care of self/family, skills building, and eating healthy; 2) Individual 1:1 weekly ASHA support; and 3) referral to grant-supported life skills classes taught by experts.
  Interventions: Behavioral: ASHA-Health HPV Intervention
- SOC+ (Other): The investigators will offer an enhanced standard of care to include usual care + three (1.5 hour) group sessions on wellness, basic nutrition, coping with mental health issues, importance of HPV screening and treatment as needed, and ART adherence (similar to Modules for ASHA-Health), and similarly delivered by the nurse and content experts over the six-month intervention.
  Interventions: Behavioral: Enhanced Standard of Care (SOC+)

INTERVENTIONS:
Behavioral: ASHA-Health HPV Intervention — The ASHA-Health HPV program will include three components: 1) Individual 1:1 weekly ASHA support; 2) 8 group sessions for the 42 W-Co-V in the ASHAHealth cohort, covering content in Modules 1-4; and 3) referral to life skills classes. The assigned ASHA will provide services to support the W-Co- V in accessing and/or adhering to HPV and ART appointments (arrange transportation, provide counseling, promote healthy lifestyle choices, and link with community resources). ASHA will also promote positive coping, social support, and aid in dealing with stigma. The 8 group sessions will be held over the six months, based on the needs identified by the women. Overall, the intervention content targets the provision of emotional support, skill building, HPV/ HIV and nutrition education, and protein-enriched food supplements, and ways to deal with stress, stigma, and the importance of engagement and retention in care. Food selections will be guided by our nutrition experts.
  Arms: ASHA-Health
Behavioral: Enhanced Standard of Care (SOC+) — Selecting our base at the Belgaum ART Centers will provide the most up to date services for the SOC+ group. Yet, there is no typical standard of care in India as it relates to HPV screening for W-Co-V and stigma associated with both diseases is high. Further, in India, screening services are lacking at most ART centers. Since it would be unethical to withhold potentially lifesaving information about HPV, the investigators will offer an enhanced standard of care to include usual care + 3 (1.5 hour) group sessions on wellness, basic nutrition, coping with mental health issues, and HIV/ HPV information. Thus, women will meet as a group three times over the six-month period. In addition, the women have access to our SOC+ nurse and ASHA to respond to questions.
  Arms: SOC+

SUMMARY:
Cervical cancer (CC) remains one of the most common malignancies among women in India, with nearly 100,000 women diagnosed annually and over 60,000 preventable deaths annually. With high-risk human papillomavirus (HR-HPV) as the causative agent for CC, one risk factor that places women at high risk for CC is human immunodeficiency virus (HIV), as impaired immune response against Human papillomavirus (HPV) may result in persistent HR-HPV infection, a critical risk factor for progression of HPV-related cervical oncogenesis. Progression of precancerous lesions among women living with HIV (WLH) is also associated with: 1) lack of HPV screening; 2) high levels of depressive symptoms and stigma; and 3) malnutrition, which negatively impacts the activation and proliferation of immune cells. Yet programs that offer WLH with comprehensive services focused on HPV screening and psychological and nutritional support are almost non-existent, and the gap is critical. Nutrition plays an integral role in relationship to HPV/HIV co-infection, as demonstrated by an increased risk of HR-HPV associated with poor nutrition; nutritional deficiencies are likewise linked to cervical intra-epithelial neoplasia. The immunological effect of malnutrition may also be exacerbated among WLH due to elevated energy demands of chronic immune activation; worsened with HPV/HIV co-infection. Further, depressive symptoms (aka depression for brevity) partially mediate the effect of food insecurity on HIV viral suppression. In our completed ASHA-Nutrition R01 study of antiretroviral (ART) adherence, the investigators trained lay community health workers, named Accredited Social Health Activist (ASHA), to improve the health of 600 rural WLH by providing emotional support, skill-building, nutrition education, and/or protein-enriched food supplements. In that study, our intervention, co-delivered by our trained ASHA, and guided by nurses, led to increased CD4+ T cell recovery and improved anthropometric and psychosocial outcomes. The investigators found that ASHA support plus protein supplements and nutritional education were significantly associated with improved CD4 counts and increased lean mass at 18 months (P < 0.001), as well as significant improvements in depression, ART adherence, social support and internalized stigma. In our sub study, CC screening of 598 of these WLH revealed that 13% were found to have abnormal cervical lesions and 4 (1%) had squamous CC. Preliminary evidence also revealed that nutritional supplements may be associated with a 40% reduction in the risk of abnormal cervical lesions (adjusted odds ratio [aOR] = 0.60), with an association between serum albumin and reduced risk of abnormal lesions (aOR= 0.39).

With a focus on secondary prevention of CC, the investigators hope to mitigate the link between HR-HPV persistence and risk of CC as well as improve the health of women co-infected with HPV/HIV (W-Co-V). Our stellar team plans to build upon our prior ASHA-Nutrition intervention, using formative research to refine a nurse-led, ASHA co-delivered, nutrition-enhanced ASHA-Health HPV intervention, adapted for W-Co-V. This will be followed by a randomized controlled trial (RCT), assessing the efficacy of our refined comprehensive, multifaceted ASHA-Health HPV intervention, as compared with an enhanced Standard of Care (SOC+) (usual care + 3 sessions [wellness, basic nutrition and HPV/HIV health promotion]) among 420 high-risk co-infected women to prevent CC while remaining engaged in the HIV treatment cascade, and managing nutritional health. Participants, recruited from a total of 24 villages, will be individually randomized in a 1:1 ratio into the two study arms. Our Primary outcome is HR-HPV persistence (2 positive tests for the same HR-HPV type, separated by 12-18 months). The two aims incorporating RCT interventions are as follows:

Aim 2. To evaluate the efficacy of ASHA-Health HPV intervention among 420 W-Co-V on the primary outcome (HR-HPV persistence) as compared to the Enhanced Standard of Care (SOC+) program. H2: Compared to the SOC+ participants, ASHA-Health participants will have lower rates of HR-HPV persistence.

Aim 3. Assess the impact of the ASHA-Health program secondarily on: 1) HIV indices (HIV viral load; CD4 count); 2) Nutritional index (serum albumin) at 6-, 12-, and 18-months.

DETAILED DESCRIPTION:
In this 5-year parallel-group RCT, the investigators will conduct a RCT to assess the efficacy of our six-month ASHA-Health HPV intervention, featuring: 1) eight in-depth group education sessions by nurses, OB/GYN and HIV physicians, psychologists, and nutrition experts on HPV/HIV, CC, and nutrition; 2) ASHA supported 1:1 sessions and community referrals; and 3) selected life skills training by expert artisans as compared to an Enhanced Standard of Care (SOC+) program, featuring 3 group sessions: wellness, basic nutrition and HIV/HPV information and referrals. The primary outcome is HR-HPV persistence (consecutive positivity for same HR-HPV type, separated by 12-18 months).

Secondary outcomes include improved: 1) HIV-related indices (HIV viral load and CD4 count); 2) Nutritional indices (serum albumin) measured at 6, 12, and 18 mos.

The investigators will conduct a two-arm parallel-group RCT among 420 W-Co-V who are cared for at the Belgaum District ART centers. Participants from 24 villages in Karnataka will be individually randomized in a 1:1 ratio to the ASHA-Health and SOC+ study arms prior to enrollment. A cohort of 84 women (42 per group) will be enrolled every six months. Primary outcome, HR-HPV persistence (positivity for same HR-HPV type, separated by 12-18 months), will be compared to enhanced standard of care (SOC+) control group that is above and beyond what is typically offered to WLH treated in the health facility. Persistent HR-HPV is a widely used outcome for HPV vaccine and other CC prevention interventions, due to its critical role in HPV-related cervical oncogenesis. Secondary outcomes will focus on improvement in: 1) HIV related indices (HIV viral load and CD4 count); and 2) Nutritional index, serum albumin levels - a marker for protein consumption).

Setting: Karnataka is selected as our key site for the study as rates of HPV have remained second highest in the country. The W-Co-V will be recruited from underserved ART centers in the Belgaum District of Karnataka which include Belgaum, Athani, Chikooi, Gokak, Raibagh and Saudatti. These ART centers are surrounded by a total of 24 villages from which approximately 17.5 women will be enrolled from each. A recent study in Delhi revealed HPV prevalence to range from 23.8% to 32.2% among WLH who attended ART clinics, while in a Mumbai-based study, HPV prevalence was 35.7% among WLH. The KSAPS (Karnataka State acquired immunodeficiency syndrome (AIDS) Program Society) has approved these sites to participate in our study and has provided demographics as follows: Across all ART sites, about 150 new WLH are enrolled each month and approximately 25% (37 per month) will be HR-HPV positive and meet other eligibility criteria. Among these 37, the investigators anticipate 50% (18-19 WLH) will be found to be negative on the visual inspection with acetic acid (VIA) of the cervix, of whom 15 new WLH would be eligible to monthly or as new cohorts are enrolled every six months; this would provide a pool of approximately 90 W-Co-V every six months. In addition, there are about 400 existing WLH who are eligible to be considered for initial assessment. To enroll 420 W-Co-V, a total of 4200 WLH will be screened; thus, ongoing screening of our staff will be conducted in all 6 ART centers. In our recently completed ASHA-Nutrition R01 study, the investigators screened 972 WLA and enrolled 600 eligible WLA; one full-time interviewer continuously screened and prepared WLH for enrollment from 45 villages (4 mandales). ASHA were also trained to assist in screening and recruitment throughout the study as there was one-month period in between cohorts to allow for ASHA support. They were also well trained to ensure accidental disclosure did not occur. In the proposed study, the investigators plan on hiring and training two full-time interviewers who will be recruiting from 24 villages, and similarly, with screening and recruitment support from ASHA, 4200 participants will be screened over 27 months. That would equate to screening 155 women each month: 77 per interviewer. Over a 20-day month, the total number of women screened can be over 100.

First-line ART is offered free by the government to all eligible PLWH and all newly diagnosed are referred to the ART centers. Thus, the investigators anticipate the 6 ART Centers will provide a sufficient number of eligible women. Screening and Enrollment Procedure: The interviewers will inform the WLH about the study with flyers posted in the lobbies of the ART centers. Interested WLH will approach the interviewer, stationed in the lobby, and retreat to a private room for further information. After the study is discussed, and all questions answered, the initial informed consent form (ICF) for screening will be signed by the WLH. Immediately thereafter, the interviewer will administer a brief 5-minute screening assessing age, prior HPV screening/treatment for HPV, abnormal cytology/CC, and HIV and ART status. Those who found not eligible will be thanked for their time, provided the screening compensation and provided any immediately needed referrals in the community. Among those eligible, HPV status will be assessed by requesting the women to perform a self-sample vaginal swab collection in their home or the nearby restroom, wherein trained ASHA will be available to assist. The samples will be collected and sent to a selected lab for processing. At the lab, the samples will be processed for presence of oncogenic HPV, and genotyping as a packaged product by Lalpathlabs, the largest lab in India. If oncogenic type HPV is found, a visual inspection of the cervix with application of acetic acid will be scheduled and conducted by our trained auxiliary nurse midwife (ANM). Typically, in India, ANMs are trained to do VIAs; a good substitute for CC screening in low resource areas. To enhance validity of interpretation and have a documentable and retrievable image of the cervix, the investigators will capture pre-VIA and post-VIA image of the cervix using a mobile app, which will be stored and interpreted by our gynecologist, along with our ANM, to enhance the accuracy of the ANM. Results will be provided confidentially to the woman by the ANM, under the guidance of protocols developed by our gynecologist. If found to be VIA negative, the W-CoV will be referred to the interviewer for consideration of enrollment into the study, and a second ICF for participating in the RCT will be discussed and signed. Women found to be VIA positive will be immediately referred to a gynecologist. Eligible and consenting women will be individually randomized in a 1:1 ratio to either the ASHA-Health or SOC+ programs prior to study initiation. Once assigned, the PC will deliver the assignment to the appropriate study nurse and ASHA.

Based on world health organization (WHO) guidelines, WLH found to be HPV positive should be rescreened for HPV in the next 12 months, along with VIA. If found to be VIA negative, screening can be resumed every 3 years. The interview staff are not involved in the delivery of the intervention and thus are blinded to condition for all assessments. Providers at the ART centers will also be blinded to study conditions.

Study Procedure: The investigators will enroll 420 eligible W-Co-V into one of two programs; cohorts of 42 WLH per program (total 84), will be initiated; each of the five program cohorts will be enrolled in the study for six months. Followup assessments will occur at 6, 12, and 18 months. New cohorts of 84 WLH (42 per program) will be enrolled upon completion of the prior six-month cohort; enrollment will be completed by month 36. For all enrolled women, the three-day, 24-hour recall (3 days prior to the baseline questionnaire administration) will be conducted. These 24 hour recalls, conducted by blinded interviewers, are designed to assess food consumption at baseline, and at all follow-ups. Also, on the 3rd day, the remaining baseline surveys will be administered by the blinded interviewer in the research office, with data entered into the tablets, inclusive of Bioelectrical Impedance Analysis (BIA) assessments. As a process measure, 24-hour recalls (1 day) will continue monthly (1-5), either just before their group session at the research office, or by home visit, by the interviewer, along with ART adherence for both groups, and at 12 and 18-month follow-ups, while the 3-day recall will be conducted just prior to baseline and again at month 6. As BIA is conducted by an office-based instrument, assessments will be conducted at baseline and months 1, 3, and 5, and at follow-up for both groups. For the study, the investigators will recruit and train 7 ASHA who reside near the targeted villages of assigned women. For the ASHA-Health group of 42 per cohort, 5 ASHA will be hired and trained. For the SOC+ group, 2 ASHA will be hired and separately trained and will support the SOC+ group. Due to differential workload, the 2 control ASHA will each be responsible for 22 SOC+ participants per cohort. To mitigate self-selection, in addition to analyzing differences between women who agree vs do not agree to participate in terms of demographics collected during screening, the interviewers and ASHA will be well trained to promote comfort and mitigate their potential fear of unwanted disclosure, as well as recruit from multiple settings and at different times of day to try to get as wide and representative range as possible.

ASHA-Health Intervention (Program 1): After the intervention ASHA have received their training, each will be assigned to their subgroup of W-Co-V to provide 1:1 support. An ASHA-Health nurse will guide the 5 ASHA; each ASHA will be assigned 8-9 women in their cohort. The ASHA will interact with their cohort weekly to assess, monitor and conduct all activities based on protocol over a six-month period. Based on an initial interview of the nurse and assigned ASHA, a needs assessment will be conducted to assess the most pressing barriers to intervention participation and completion, and the tailored assessment will be integrated into the unique plan for each participant. Nevertheless, the major components of the program will be delivered to all women assigned to that program. To address these general needs reported by the nearly 600 WLH regarding CC screening in our ASHA-Nutrition program, the ASHA-Health program will include: 1) 8 group sessions, led by the nurse, and inclusive of other experts (such as HPV/HIV physician, nutritionist, psychologist) to provide the group classes for each cohort of 42 W-Co-V in the program, covering content in Modules 1-4; 2) Individual 1:1 weekly ASHA support; and 3) referral to grant-supported life skills classes taught by experts.

The specific classes relevant to our targeted W-Co-V will be assessed in our CAB/focus group discussions, but might include selling vegetables, sewing, weaving, embroidery, etc. These classes will provide economic sustainability, as accomplished by 80% of the WLH in our ASHA-Nutrition study. In the 8 group sessions, based on the comprehensive health seeking and coping paradigm (CHSCP), the nurse and content experts in Nursing, Medicine, Psychology and Nutrition will address distinct barriers to ongoing engagement in care by educating the cohort about health promotion, HPV/HIV, coping with stigma, improving depressive symptoms, seeking trusted supports, and keeping mentally healthy. The ASHA who cares for these women will also attend, listen to the program, and support the team. The assigned ASHA will make weekly home visits and focus on providing 1:1 support to the W-Co-V in accessing and/or adhering to ART as well as reinforcing education received in group sessions, assisting with transportation, offering to accompany them to appointments, providing counseling, promote healthy lifestyle choices, and links with community resources. This weekly ASHA support will occur over the six-month intervention. Records of time spent will be carefully monitored on the tablets. As lack of job skills has been previously identified as a source of stress, the ASHA will assess job skills of interest for each woman and arrange selected training sessions weekly over the six-month period with skilled artisans. The 8 (1.5 hours) group sessions will be held bimonthly over the first four months in a space the research team will rent that is central to all villages, based on the needs identified by prior WLH, and updated by the planned community advisory board (CAB), focus group (FG) meetings, and needs assessment. In months 5 and 6 of the program, the ASHA will hold role play sessions once a month where the cohort will come together, and role play what they have learned in group sessions and how they are implementing it. Module 1 (sessions 1 & 2) will provide general information on HPV, the importance of seeking support from ASHA, healthcare providers and trusted family/friends; importance of routine HPV screening per WHO guidelines after being diagnosed as HPV+, ART adherence, basics of nutrition, and keeping healthy routines, such as immune strengthening diet, adequate rest, etc. Module 2 (sessions 3 & 4) will focus on caring for self and family, in-depth discussion of CC, and HPV screening, discussions by experts on ways to enhance coping, including legal and spiritual; and beginning life skills vocational classes. In Module 3 (sessions 5 & 6), the focus will be skills building, strategies to improve coping, stigma and problem solving, all of which will build resilience; pros and cons of disclosure; continued life skills, and ways to increase community awareness of HPV. Module 4 (sessions 7 & 8) will focus on providing education about which foods are the least expensive, easily accessible, and highly nutritious and immune supportive; and sharing recipes and enjoying cooking classes. Our nutrition experts will guide food selections using the Dietary Guidelines for Indians and food availability in the local region. Finally, ASHA will provide monthly food supplements that will consist of high protein foods (i.e. Dal lentils), while attending to minimal saturated fat, fiber (soluble fiber), and the cholesterol content of the foods. Food will be distributed based on family size with enough food for each family member to ensure the participant receives the intervention. In addition, to accommodate women who are unable to make group-assigned classes, additional flexible dates will be offered. If successful, this intervention can be easily scaled up by integrating ASHA training into the current Health Mission of India strategies.

Enhanced Standard of Care (SOC+): In India, screening services are lacking at most ART centers. Since it would be unethical to withhold potentially lifesaving information about HPV, the investigators will offer an enhanced standard of care to include usual care + three (1.5 hour) group sessions on wellness, basic nutrition, coping with mental health issues, importance of HPV screening and treatment as needed, and ART adherence, and similarly delivered by the nurse and content experts over the six-month intervention. Women assigned to the SOC+ program will be HPV screened at baseline as well and will meet as a group three times to meet their distinct SOC+ nurse and ASHA at the research site. The SOC+ nurse and ASHA, trained separately from the ASHA-Health nurse and ASHA, will provide information on resources in the community, including nutritious and low-cost foods, as well as referral to ART and other services as needed, and remind the participants by phone of upcoming appointments. However, ASHA will not be visiting the women in their homes, nor will they receive the other modules or food supplements. Each of the two SOC+ ASHA will follow their cohort of 22 participants over the six-month period. The SOC+ nurse will guide their ASHA and answer medical questions for their participants.

ELIGIBILITY:
Inclusion Criteria:

1. WLH, 25 - 50 years of age; based on HIV-based guidelines;
2. Receiving ART for > 12 months to ensure medication stabilization, and ensure any impact on the cervical cancer outcomes will not be attributed solely to recent ART initiation, as validated by an ART card given to all ART patients;
3. Screened as HPV positive by RT-PCR (Reverse Transcription Polymerase Chain Reaction) for oncogenic genes; and assessed to be VIA negative;
4. Have not participated in Phase I Formative Study.

Exclusion Criteria:

1. Pregnant or lactating women due to hormonal and dietary guideline differences;
2. Women older than age 50. These women will be immediately referred to a gynecology specialist.

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 420 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
HR-HPV Detection | Baseline and month 6, 12 and 18 month follow-ups
  HR- HPV test will detect 14 oncogenic HR-HPV genotypes (HPV16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68). HR-HPV persistence is defined as the presence of the same genotype over at least 12 months.

SECONDARY OUTCOMES:
HIV Viral Load | Baseline and month 6, 12, and 18
  The investigators will measure HIV viral load using the cobas TaqMan HIV-1 Test (Roche, Basel, Switzerland). HIV VL is conducted free at all ART Centers.
CD4 Count | Baseline and month 6, 12, and 18
  Will be assessed every six months and processed in real time at the clinic by flow cytometry. CD4 count has been shown to be a good predictor of various cervical outcomes. CD4 counts are conducted free at all ART Centers.
Serum-based Albumin | Baseline and month 6, 12, and 18
  Serum albumin will be collected through blood draws occurring at baseline, and 6, 12, and 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Adey Nyamathi, ANP, PhD, FAAN, Principal Investigator — UCI Sue & Bill Gross School of Nursing
Locations (1):
- KC General Hospital, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
The data will be all collected in India and Indian law prohibits sharing of individual participants' research data data with other investigators.

REFERENCES:
- [Background] Nyamathi A, Hanson AY, Salem BE, Sinha S, Ganguly KK, Leake B, Yadav K, Marfisee M. Impact of a rural village women (Asha) intervention on adherence to antiretroviral therapy in southern India. Nurs Res. 2012 Sep-Oct;61(5):353-62. doi: 10.1097/NNR.0b013e31825fe3ef. PMID 22872107
- [Background] Nyamathi A, Ekstrand M, Salem BE, Sinha S, Ganguly KK, Leake B. Impact of Asha intervention on stigma among rural Indian women with AIDS. West J Nurs Res. 2013 Aug;35(7):867-83. doi: 10.1177/0193945913482050. Epub 2013 Mar 27. PMID 23539322
- [Background] Garfin DR, Shin SS, Ekstrand ML, Yadav K, Carpenter CL, Sinha S, Nyamathi AM. Depression, social support, and stigma as predictors of quality of life over time: results from an Asha-based HIV/AIDS intervention in India. AIDS Care. 2019 May;31(5):563-571. doi: 10.1080/09540121.2018.1563281. Epub 2019 Feb 3. PMID 30714386
- [Background] Nyamathi A, Ekstrand M, Srivastava N, Carpenter CL, Salem BE, Al-Harrasi S, Ramakrishnan P, Sinha S. ASHA-Life Intervention Perspectives Voiced by Rural Indian Women Living With AIDS. Health Care Women Int. 2016;37(4):412-25. doi: 10.1080/07399332.2015.1066790. Epub 2015 Jul 6. PMID 26147930